CLINICAL TRIAL: NCT03964220
Title: The Effectiveness of Tiotropium Add-on Therapy Using a Real-world Cohort of Patients With Asthma
Brief Title: Impact of Tiotropium Add-on Therapy in Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0205-0543
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Asthma
  Interventions: Drug: Tiotropium Respimat®; Drug: Inhaled Corticosteroid/Long-acting beta-agonist

INTERVENTIONS:
Drug: Tiotropium Respimat® — Tiotropium Respimat® 1.25 mcg (on top of baseline Inhaled Corticosteroid/Long-acting beta-agonist )
Drug: Inhaled Corticosteroid/Long-acting beta-agonist — baseline low dose to medium/high dose, baseline medium dose ICS/LABA to high dose ICS/LABA, additional prescription/refill of high-dose-ICS/LABA following the first prescription of baseline high dose ICS/LABA

SUMMARY:
To evaluate the effectiveness of add on therapy with Tiotropium Respimat® compared to increasing the dose of ICS in patients with a diagnosis of Asthma and on ICS/LABA therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with least one asthma diagnosis in the inpatient setting or at least two separate instances of asthma diagnosis (separated by at least 30 days) recorded in the outpatient or emergency room setting will be included.
* Patients will be required to be already on Inhaled Corticosteroid/Long-acting beta-agonist (ICS/LABA).
* Patients will be required to have available records 12 months prior to the index date.

Exclusion Criteria:

* Patients below the age of 6 years on the Inhaled Corticosteroid/Long-acting beta-agonist initiation (ICS/LABAi) date will be excluded.
* Patients with a diagnosis of COPD at any time during the study period will be excluded.
* Those who are on biologics at baseline will be removed.
* After the PSM process, unmatched patients will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asthmatics 6 years and above on ICS/LABA at baselineIMS Pharmetrics (IMS or Database I); EMRClaims+ (Database II)
Sampling Method: Non-Probability Sample
Enrollment: 7857 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- eMax Health, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https:// trials.boehringer-ingelheim.com/trial_results/ clinical_submission_documents.html to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link http://trials.boehringeringelheim. com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://trials.boehringer-ingelheim.com

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective cohort data analysis evaluated the effectiveness of add on therapy with Tiotropium Respimat® 1.25 microgram comparing to increasing the dose of Inhaled Corticosteroid (ICS) in patients with a diagnosis of Asthma and on ICS/Long-acting beta-agonist (LABA) therapy.
Pre-assignment Details: This study included asthma patients from two retrospective data sources (IMS Pharmetrics and EMRClaims+) after propensity score matching based on ICS/LABA dose on initiation date, demographics, Charlson Comorbidity index (CCI) score, specific comorbidities, medications and asthma control status.
Groups:
- Tiotropium Respimat® (Tio Group): 1.25 microgram (mcg) of solution of inhalation of Tiotropium Respimat® added-on to Inhaled Corticosteroid (ICS)/long-acting beta-agonists (LABA) therapy.
  Advair Diskus, Advair HFA, AirDuo, Breo, Dulera or Symbicort were used for the ICS/LABA therapy from low dose (Advair Diskus (100mcg), Advair HFA (45mcg), AirDuo (55mcg), Breo (100mcg), Dulera (100mcg), Symbicort (80mcg)), to medium dose (Advair Diskus (250mcg), Advair HFA (115mcg), AirDuo (113mcg)) and high dose (Advair Diskus (500mcg), Advair HFA (230mcg), AirDuo (232mcg), Breo (200mcg), Dulera (200mcg), Symbicort (160mcg)).
- Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group): Low dose ICS/LABA to medium/high dose ICS/LABA or from baseline medium dose ICS/LABA to high dose ICS/LABA or an additional prescription/refill of high-dose ICS/LABA following the first prescription of baseline high dose ICS/LABA within the study period.
  Advair Diskus, Advair HFA, AirDuo, Breo, Dulera or Symbicort were used for the ICS/LABA therapy from low dose (Advair Diskus (100mcg), Advair HFA (45mcg), AirDuo (55mcg), Breo (100mcg), Dulera (100mcg), Symbicort (80mcg)), to medium dose (Advair Diskus (250mcg), Advair HFA (115mcg), AirDuo (113mcg)) and high dose (Advair Diskus (500mcg), Advair HFA (230mcg), AirDuo (232mcg), Breo (200mcg), Dulera (200mcg), Symbicort (160mcg)).
Period: Overall Study
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Started | 2619 | 5238
Completed | 2619 | 5238
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study included asthma patients from two retrospective data sources (IMS Pharmetrics and EMRClaims+) after propensity score matching based on ICS/LABA dose on initiation date, demographics, Charlson Comorbidity index (CCI) score, specific comorbidities, medications and asthma control status.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group) | Total
Number analyzed (Participants) | 2619 | 5238 | 7857
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.12 (15.38) | 44.77 (15.43) | 44.89 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1802 | 3576 | 5378
  Male | 817 | 1662 | 2479
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to First Exacerbation
Description: Exacerbations will be defined as either a hospitalization with a primary diagnosis of asthma, an emergency room (ER) visit with a primary diagnosis of asthma, an asthma exacerbation diagnosis recorded.
Time Frame: From baseline until end of follow-up, up to 3 years
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Number analyzed (Participants) | 2619 | 5238
Days | 340.656 (428.061) | 123.151 (152.600)
Statistical Analysis 1: Comparison: Tiotropium Respimat® (Tio Group) vs Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group); The time to first exacerbation was analysis using Cox Proportional Hazards model with group status as the only independent variable assessing the risk of exacerbation across Tio and NonTio groups; Test type: Other; p = 0.044, Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.427 to 0.990]

2. Secondary Outcome: Rate of Exacerbation at 6 Months and 1 Year of Follow-up
Description: Exacerbation rate per 100 person-years. Follow-up period was from index date (date of the first prescription for Tiotropium Respimat® 1.25 mcg in Tio group; date of the first prescription from low to medium/high does or medium to high does or additional high-does of Inhaled Corticosteroid (ICS)/long-acting beta-agonists (LABA) for NonTio group).
Time Frame: At 6 month and 1 year of follow-up
Population: as for baseline characteristics
Measure: Number; unit: Events per 100 person-years
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Number analyzed (Participants) | 2619 | 5238
Events per 100 person-years
  At 6 months of follow-up | 41.40 | 116.07
  At 1 year of follow-up | 15.65 | 57.24
Statistical Analysis 1: Comparison: Tiotropium Respimat® (Tio Group) vs Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group); Analysis for the rate of exacerbation between Tio and NonTio groups within 6 months of follow-up; Test type: Other; p < 0.0001, Negative binomial regression
Statistical Analysis 2: Comparison: Tiotropium Respimat® (Tio Group) vs Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group); Analysis for the rate of exacerbation between Tio and NonTio groups within 1 year of follow-up; Test type: Other; p < 0.0001, Negative binomial regression

3. Secondary Outcome: Health Care Resource Utilization (HCRU) During Follow-up
Description: Follow-up period was from index date (date of the first prescription for Tiotropium Respimat® 1.25 mcg in Tio group; date of the first prescription from low to medium/high does or medium to high does or additional high-does of Inhaled Corticosteroid (ICS)/long-acting beta-agonists (LABA) for NonTio group) and up to 3 years of study period.
Time Frame: During follow-up period, From baseline until end of follow-up, up to 3 years
Population: as for baseline characteristics
Measure: Number; unit: Events per 100 person-years
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Number analyzed (Participants) | 2619 | 5238
Events per 100 person-years
  Hospitalization (all cause) | 23.97 | 46.51
  Hospitalization (asthma related) | 4.89 | 20.27
  Emergency room (ER) visit (all cause) | 45.00 | 84.67
  ER visit (asthma related) | 12.23 | 47.70
  Outpatient (OP) visit (all cause) | 206.92 | 232.55
  OP visit (asthma related) | 133.06 | 158.61

4. Secondary Outcome: Change in Lung Function (Forced Expiratory Volume in 1 Second (FEV1) Score) at Baseline and Follow up Period
Description: Follow-up period was from index date (date of the first prescription for Tiotropium Respimat® 1.25 mcg in Tio group; date of the first prescription from low to medium/high does or medium to high does or additional high-does of Inhaled Corticosteroid (ICS)/long-acting beta-agonists (LABA) for NonTio group) and up to 3 years of study period. FEV1 score range from 0 to 100. Higher FEV1 score suggests normal lung function, while lower for dangerous. Only the descriptive statistics of FEV1 score were reported other than change of FEV1 score from baseline due to lack of enough data points.
Time Frame: From baseline until end of follow-up, up to 3 years
Population: This study included asthma patients from two retrospective data sources (IMS Pharmetrics and EMRClaims+) after propensity score matching based on ICS/LABA dose on initiation date, demographics, CCI score, specific comorbidities, medications and asthma control status. Analysis conducted with participants with non-missing endpoint results.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Number analyzed (Participants) | 13 | 26
Score on a scale | 77.77 (20.16) | 85.69 (20.77)

5. Secondary Outcome: Change in Asthma Control Test (ACT) Score at Baseline and in the Follow up Period
Description: Follow-up period was from index date (date of the first prescription for Tiotropium Respimat® 1.25 mcg in Tio group; date of the first prescription from low to medium/high does or medium to high does or additional high-does of Inhaled Corticosteroid (ICS)/long-acting beta-agonists (LABA) for NonTio group) and up to 3 years of study period. ACT score is based on a range of 5 to 25. Higher score indicates better asthma control. A score of 19 or less may be a sign that asthma symptoms not under control. Only the descriptive statistics of ACT score were reported other than change of ACT score from baseline due to lack of enough data points.
Time Frame: From baseline until end of follow-up, up to 3 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
Number analyzed (Participants) | 23 | 31
Score on a scale | 15.65 (7.0) | 16.16 (5.3)

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study
Description: As this is a non-interventional study with secondary use of data retrieved from IMS Pharmetrics and EMRClaims+® database, safety monitoring and safety reporting on an individual case level is not applicable.
Arm/Group | Tiotropium Respimat® (Tio Group) | Inhaled Corticosteroid/Long-acting Beta-agonist (NonTio Group)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03964220/Prot_SAP_000.pdf